CLINICAL TRIAL: NCT07346872
Title: Comparison of EXORA Block and Epidural Analgesia on Quality of Recovery and Postoperative Analgesia Following Gynecological Surgery
Brief Title: EXORA Block vs Epidural Analgesia in Gynecological Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BursaYIEAH-2024
Record Dates: First submitted 2025-12-28; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pain; Postoperative Pain
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Tramadol; Injections, Epidural

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group : exora block (Active Comparator): Patients will receive an ultrasound-guided EXORA block for postoperative analgesia, performed by the attending anesthesiologist according to institutional clinical practice.
  Interventions: Drug: Tramadol; Procedure: exora block
- Group:Epidural Analgesia (Active Comparator): Patients will receive epidural analgesia for postoperative pain control, administered by the attending anesthesiologist according to standard institutional protocols.
  Interventions: Drug: Tramadol; Procedure: epidural

INTERVENTIONS:
Drug: Tramadol — 400 mg tramadol, IV 4 mg/ mL tramadol solution into 100 mL normal saline; Patient-controlled analgesia settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
Procedure: exora block — Ultrasound guided External Oblique And Rectus Abdominis Plane (EXORA) Block block (0.3 ml/kg , %0.25 bupivacaine) will be performed
  Arms: Group : exora block
Procedure: epidural — Thoracic epidural catheterization will be performed preoperatively at the Thoracic 8-Thoracic 10 levels. Postoperatively, a bolus dose of 10 ml of 0.25% local anesthetic will be administered followed by continuous infusion.
  Arms: Group:Epidural Analgesia

SUMMARY:
This prospective observational study aims to compare the effects of the EXORA block and epidural analgesia on postoperative pain control and quality of recovery in patients undergoing gynecological surgery. Quality of recovery will be assessed using the Quality of Recovery-15 (QoR-15) questionnaire, and postoperative pain will be evaluated using the Visual Analog Scale (VAS).

DETAILED DESCRIPTION:
Effective postoperative analgesia is essential for improving recovery quality and patient satisfaction following gynecological surgery. Epidural analgesia is widely accepted as a standard technique for postoperative pain control; however, it may be associated with adverse effects such as hypotension and delayed mobilization. The EXORA block is an ultrasound-guided fascial plane block that has recently emerged as an alternative analgesic technique with a potentially favorable safety and recovery profile.

This prospective observational study compares postoperative recovery quality and analgesic efficacy between patients receiving EXORA block and those receiving epidural analgesia for postoperative pain management. Recovery quality will be objectively evaluated using the validated Quality of Recovery-15 (QoR-15) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 years
* ASA (American Society of Anaesthetists) physical status classification I-III
* Undergoing elective gynecological surgery
* Receiving either EXORA block or epidural analgesia for postoperative pain management

Exclusion Criteria:

* Secondary or repeat surgical procedures
* Severe renal or hepatic dysfunction
* Body mass index (BMI) greater than 30 kg/m²
* Psychiatric or cognitive disorders impairing cooperation or questionnaire completion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
NRS | Postoperative 24 hours
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

SECONDARY OUTCOMES:
Quality of Recovery-15 (QoR-15) Score | Postoperative 24 hours
  The QoR-15 is a reliable and validated tool for assessing patient-reported postoperative recovery and provides a comprehensive evaluation of physical and emotional well-being after surgery.
Total Postoperative Tramadol Consumption (mg) | Postoperative 24 hours]
  Total amount of tramadol administered for postoperative analgesia will be recorded in milligrams during the first 24 hours after surgery.
Incidence and Severity of Postoperative Nausea and Vomiting Assessed by the Nausea and Vomiting Scale (NVS) | Postoperative 24 hours
  Postoperative nausea and vomiting will be assessed using the Nausea and Vomiting Scale (NVS), defined as:
  0 = No nausea
  1. = Mild nausea
  2. = Severe nausea
  3. = Vomiting
  In cases of an NVS score ≥3, an antiemetic drug will be administered.
Number of Participants Requiring Additional Postoperative Rescue Analgesia | postoperative 24 hour
  The number of participants requiring additional postoperative rescue analgesia beyond the standard analgesic protocol within the first 24 hours after surgery will be recorded.
pinprick test | postoperative 24 hour
  The level of sensory block will be evaluated by pinprick test at 30 minutes following the block procedure and in postoperative patients.
  With the pinprick, the gently touches the skin with the pin or back end and asks the patient whether it feels sharp or blunt.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Korgün Ökmen, Bursa
  - University of Health Sciences,,Bursa Yuksek Ihtisas Training and Research Hospital,, Bursa